CLINICAL TRIAL: NCT04880603
Title: Utility of Restrata With Split-thickness Skin Graft to Reconstruct the Forearm Donor Site
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigators no longer interested in pursuing
Sponsor: Nebraska Methodist Health System (Other)
Collaborators: Acera Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Restrata
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- A - Standard of Care (Active Comparator)
  Interventions: Procedure: Standard of Care Skin Graft
- B - Restrata Graft (Experimental)
  Interventions: Device: Restrata Graft

INTERVENTIONS:
Device: Restrata Graft — Restrata will be meshed in a 1:2 fashion to allow for egress of serous fluid and minimize risk of fluid collection. Restrata will be applied to the entire wound bed not amenable to primary closure and will be underlaid beneath the surrounding skin edges. A split-thickness skin graft is harvested from patient's thigh at 15:1000 inches and placed on top of the Restrata to cover the entire wound bed. The graft is sutured in place using suture choice of surgeon's preference.
  Arms: B - Restrata Graft
Procedure: Standard of Care Skin Graft — Standard of Care Skin Graft
  Arms: A - Standard of Care

SUMMARY:
Adult patients undergoing a radial forearm free flap or ulnar forearm free flap will be randomized to the use of the Restrata graft in combination with split-thickness skin graft for reconstruction. Photos will document whether the Restata graft aids in the healing.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 19 or greater that will undergo radial forearm free flap or ulnar free flap.
* Photo documentation of wound bed at two weeks and four weeks must be obtainable either by physician or patient.

Exclusion Criteria:

* Active systemic immunosuppression (active use of high-dose steroids (≥40mg prednisone daily or equivalent) or other immunosuppressive medications OR medical conditions causing immunosuppression, i.e. human immunodeficiency virus etc).
* Diabetes mellitus with most recent Hemoglobin A1c ≥10.0 within 30 days prior to surgery.
* Morbid obesity (BMI >40).
* Inability to maintain wrist immobilization for full planned period.
* Severe malnutrition (prealbumin levels <10 mg per dL within 30 days prior to surgery OR BMI <15 (very severely underweight).
* Other conditions felt to significantly impair wound healing per surgeon discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Tendon exposure | 4 weeks post-operation
  Tendon exposure at four weeks post-operatively (Yes/No).
Percentage of surface area | 4 weeks post operation
  Percentage of surface area of split-thickness skin graft incorporation at four weeks postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lindau, MD, Principal Investigator — Nebraska Methodist Hospital
Locations (1):
- Nebraska Methodist Hospital, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No